CLINICAL TRIAL: NCT00722527
Title: Molecular Biology of Polycythemia and Thrombocytosis
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17665; 5R01HL050077-13 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Polycythemia; Thrombocytosis
Keywords: Primary Familial and Congenital Polycythemia; Polycythemia; Molecular Biology; Genetics; Erythropoiesis; EPOR mutation; Thrombocytosis; Hypoxia
MeSH Terms: conditions — Polycythemia; Thrombocytosis; Polycythemia, primary familial and congenital; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Affected Population: Subjects with an elevated hemoglobin concentration or an elevated platelet count

SUMMARY:
Our study is designed to characterize the clinical picture and genetic pattern of Polycythemia and Thrombocytosis. The purpose of this project is to find a gene and its mutation that causes these disorders. When this is accomplished, new therapies to control and eventually cure the disorder can be designed.

DETAILED DESCRIPTION:
Our hypothesis is that genes and their mutation are causative of certain types of polycythemia and thrombocytosis. These will be sought for by genetic and cell biology means. The purpose of the study is to identify the molecular defect of these disorders.

5-7 teaspoons of peripheral blood will be drawn on all study subjects. After DNA is obtained, linkage analysis and/or mutation analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with an elevated hemoglobin concentration (>18 in males and >16 in females)
2. Subjects with an elevated platelet count (>450,000)

Exclusion Criteria:

1. Subjects who have a known acquired cause of polycythemia and thrombocytosis
2. Subjects with heart disease, left to right heart shunt or severe pulmonary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have polycythemia and thrombocytosis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-07; Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Identify the molecular defect of Polycythemic and Thrombocythemic disorders | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Josef T. Prchal, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Percy MJ, Sanchez M, Swierczek S, McMullin MF, Mojica-Henshaw MP, Muckenthaler MU, Prchal JT, Hentze MW. Is congenital secondary erythrocytosis/polycythemia caused by activating mutations within the HIF-2 alpha iron-responsive element? Blood. 2007 Oct 1;110(7):2776-7. doi: 10.1182/blood-2007-03-082503. No abstract available. PMID 17881647
- [Background] Skoda R, Prchal JT. Lessons from familial myeloproliferative disorders. Semin Hematol. 2005 Oct;42(4):266-73. doi: 10.1053/j.seminhematol.2005.08.002. PMID 16210040
- [Background] Gregg XT, Prchal JT. Recent advances in the molecular biology of congenital polycythemias and polycythemia vera. Curr Hematol Rep. 2005 May;4(3):238-42. PMID 15865879
- [Background] Bento MC, Chang KT, Guan Y, Liu E, Caldas G, Gatti RA, Prchal JT. Congenital polycythemia with homozygous and heterozygous mutations of von Hippel-Lindau gene: five new Caucasian patients. Haematologica. 2005 Jan;90(1):128-9. PMID 15642680
- [Background] Jedlickova K, Stockton DW, Prchal JT. Possible primary familial and congenital polycythemia locus at 7q22.1-7q22.2. Blood Cells Mol Dis. 2003 Nov-Dec;31(3):327-31. doi: 10.1016/s1079-9796(03)00167-0. PMID 14636647
- [Result] Prchal JT, Gordeuk VR. The HIF2A gene in familial erythrocytosis. N Engl J Med. 2008 May 1;358(18):1966; author reply 1966-7. No abstract available. PMID 18456917
- [Result] Agarwal N, Mojica-Henshaw MP, Simmons ED, Hussey D, Ou CN, Prchal JT. Familial polycythemia caused by a novel mutation in the beta globin gene: essential role of P50 in evaluation of familial polycythemia. Int J Med Sci. 2007 Oct 4;4(4):232-6. doi: 10.7150/ijms.4.232. PMID 17952198